CLINICAL TRIAL: NCT01864603
Title: Sustainable East Africa Research in Community Health
Acronym: SEARCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other); Kenya Medical Research Institute (Other); Gilead Sciences (Industry); World Bank (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); United States President's Emergency Plan for AIDS Relief (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SEARCH
Record Dates: First submitted 2013-04-26; First posted 2013-05-29 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: HIV; Tuberculosis; Hypertension; Diabetes; Maternal Child Health; Cost Effectiveness
Keywords: HIV treatment and prevention; Tuberculosis; Community health campaign; PrEP
MeSH Terms: conditions — Tuberculosis; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1st: universal test and treat; 2nd: targeted PrEP and cascade (Experimental): Intervention arm first phase: annual universal community-based HIV and multi-disease testing; ART for all HIV+ using streamlined care delivery
  Intervention arm second phase: baseline universal community-based HIV and multi-disease testing; ART for all HIV+ using streamlined care delivery + targeted PrEP, and targeted HIV testing interventions
  Interventions: Other: Universal ART in a streamlined care model; Other: Annual Community Health Campaigns; Other: Targeted PrEP and Targeted testing interventions
- 1st: baseline community testing; 2nd: None (Active Comparator): Comparator arm first phase: baseline community-based HIV and multi-disease testing; ART by country standard of care
  Interventions: Other: Universal ART in a streamlined care model; Other: Baseline community-based HIV and multi-disease testing

INTERVENTIONS:
Other: Universal ART in a streamlined care model — immediate ART start for all HIV+ in community with streamlined care
Other: Annual Community Health Campaigns — HIV and multi-disease testing for all community members
  Arms: 1st: universal test and treat; 2nd: targeted PrEP and cascade
Other: Targeted PrEP and Targeted testing interventions
  Arms: 1st: universal test and treat; 2nd: targeted PrEP and cascade
Other: Baseline community-based HIV and multi-disease testing — HIV and multi-disease testing for all community members at baseline only
  Arms: 1st: baseline community testing; 2nd: None

SUMMARY:
The SEARCH study aims to test evidenced-based innovative community based interventions that lead to the elimination of HIV in rural communities in East Africa using a multi-disease approach. The first phase of the study will quantify the impact of early HIV diagnosis using a streamlined and immediate ART (antiretroviral therapy). The second phase of the study, will quantify the impact of targeted Pre-Exposure Prophylaxis (PrEP) in the context of universal treatment and streamlined care. The study intervention is designed to improve the entire continuum of care, to reduce structural barriers for all populations including those most "at risk".

DETAILED DESCRIPTION:
The SEARCH study aims to test evidenced-based innovative community based interventions that lead to the elimination of HIV in rural communities in East Africa using a multi-disease approach. The first phase of the study will quantify the impact of early HIV diagnosis using a streamlined and immediate ART (antiretroviral therapy). The second phase of the study, will quantify the impact of targeted Pre-Exposure Prophylaxis (PrEP) in the context of universal treatment and streamlined care. The study intervention is designed to improve the entire continuum of care, to reduce structural barriers for all populations including those most "at risk".

ELIGIBILITY:
Community Level Inclusion Criteria:

* Non-adjacent geopolitical units in south-western and eastern Uganda and western Kenya.
* Most recent census population between 9,000 and 11,000 individuals.
* Served by an ART providing health center.
* Community leader commitment for study participation and implementation.
* Accessibility to health center via a maintained transportation route.
* Community location with sufficient distance from other potential study communities to limit contamination of intervention or control conditions (buffer zone)

Individual Level Inclusion Criteria:

* Residency of individual in community, defined as present in household for at least 6 months of the calendar year.

Community Level Exclusion Criteria:

* Presence of ongoing community-based ART intervention strategies that provide treatment outside of the current in-country treatment guidelines.
* An urban setting defined as a city with a population of 100,000 or more inhabitants.
* Absence of a health center able to provide ART.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150395 (Actual)
Dates: Start 2013-04; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Study Chair — University of California, San Francisco; Moses Kamya, MBChB, PhD, Principal Investigator — Makerere University; Maya Petersen, PhD, Principal Investigator — University of California, Berkeley
Locations (3):
- Nyanza Province Kenya, Nyanza Province, Kenya
- Uganda (2):
  - Eastern Uganda, Mbale/Tororo Region
  - Southwestern Uganda, Mbarara Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balzer LB, Petersen ML, van der Laan MJ; SEARCH Consortium. Adaptive pair-matching in randomized trials with unbiased and efficient effect estimation. Stat Med. 2015 Mar 15;34(6):999-1011. doi: 10.1002/sim.6380. Epub 2014 Nov 25. PMID 25421503
- [Background] Camlin CS, Seeley J, Viljoen L, Vernooij E, Simwinga M, Reynolds L, Reis R, Plank R, Orne-Gliemann J, McGrath N, Larmarange J, Hoddinott G, Getahun M, Charlebois ED, Bond V. Strengthening universal HIV 'test-and-treat' approaches with social science research. AIDS. 2016 Mar 27;30(6):969-70. doi: 10.1097/QAD.0000000000001008. No abstract available. PMID 26959355
- [Background] SEARCH Collaboration. Evaluating the feasibility and uptake of a community-led HIV testing and multi-disease health campaign in rural Uganda. J Int AIDS Soc. 2017 Mar 30;20(1):21514. doi: 10.7448/IAS.20.1.21514. PMID 28406269
- [Background] Balzer LB, van der Laan MJ, Petersen ML; SEARCH Collaboration. Adaptive pre-specification in randomized trials with and without pair-matching. Stat Med. 2016 Nov 10;35(25):4528-4545. doi: 10.1002/sim.7023. Epub 2016 Jul 19. PMID 27436797
- [Background] Balzer L, Staples P, Onnela JP, DeGruttola V. Using a network-based approach and targeted maximum likelihood estimation to evaluate the effect of adding pre-exposure prophylaxis to an ongoing test-and-treat trial. Clin Trials. 2017 Apr;14(2):201-210. doi: 10.1177/1740774516679666. Epub 2017 Jan 26. PMID 28124579
- [Background] Tram KH, Mwangwa F, Atukunda M, Owaraganise A, Ayieko J, Plenty A, Kwariisima D, Clark TD, Petersen ML, Charlebois ED, Kamya MR, Chamie G, Havlir DV, Marquez C; SEARCH Collaboration. Isoniazid Preventive Therapy Completion in the Era of Differentiated HIV Care. J Acquir Immune Defic Syndr. 2017 Dec 15;76(5):e115-e117. doi: 10.1097/QAI.0000000000001540. No abstract available. PMID 28885271
- [Background] Puryear SB, Balzer LB, Ayieko J, Kwarisiima D, Hahn JA, Charlebois ED, Clark TD, Cohen CR, Bukusi EA, Kamya MR, Petersen ML, Havlir DV, Chamie G. Associations between alcohol use and HIV care cascade outcomes among adults undergoing population-based HIV testing in East Africa. AIDS. 2020 Mar 1;34(3):405-413. doi: 10.1097/QAD.0000000000002427. PMID 31725431
- [Background] Balzer LB, Havlir DV, Kamya MR, Chamie G, Charlebois ED, Clark TD, Koss CA, Kwarisiima D, Ayieko J, Sang N, Kabami J, Atukunda M, Jain V, Camlin CS, Cohen CR, Bukusi EA, Van Der Laan M, Petersen ML. Machine Learning to Identify Persons at High-Risk of Human Immunodeficiency Virus Acquisition in Rural Kenya and Uganda. Clin Infect Dis. 2020 Dec 3;71(9):2326-2333. doi: 10.1093/cid/ciz1096. PMID 31697383
- [Background] Marcus JL, Sewell WC, Balzer LB, Krakower DS. Artificial Intelligence and Machine Learning for HIV Prevention: Emerging Approaches to Ending the Epidemic. Curr HIV/AIDS Rep. 2020 Jun;17(3):171-179. doi: 10.1007/s11904-020-00490-6. PMID 32347446
- [Background] Balzer LB, Ayieko J, Kwarisiima D, Chamie G, Charlebois ED, Schwab J, van der Laan MJ, Kamya MR, Havlir DV, Petersen ML. Far from MCAR: Obtaining Population-level Estimates of HIV Viral Suppression. Epidemiology. 2020 Sep;31(5):620-627. doi: 10.1097/EDE.0000000000001215. PMID 32452912
- [Background] Jewell BL, Balzer LB, Clark TD, Charlebois ED, Kwarisiima D, Kamya MR, Havlir DV, Petersen ML, Bershteyn A. Predicting HIV Incidence in the SEARCH Trial: A Mathematical Modeling Study. J Acquir Immune Defic Syndr. 2021 Aug 1;87(4):1024-1031. doi: 10.1097/QAI.0000000000002684. PMID 33770065
- [Result] Chamie G, Kwarisiima D, Clark TD, Kabami J, Jain V, Geng E, Petersen ML, Thirumurthy H, Kamya MR, Havlir DV, Charlebois ED; SEARCH Collaboration. Leveraging rapid community-based HIV testing campaigns for non-communicable diseases in rural Uganda. PLoS One. 2012;7(8):e43400. doi: 10.1371/journal.pone.0043400. Epub 2012 Aug 20. PMID 22916256
- [Result] Thirumurthy H, Chamie G, Jain V, Kabami J, Kwarisiima D, Clark TD, Geng E, Petersen ML, Charlebois ED, Kamya MR, Havlir DV; SEARCH Collaboration. Improved employment and education outcomes in households of HIV-infected adults with high CD4 cell counts: evidence from a community health campaign in Uganda. AIDS. 2013 Feb 20;27(4):627-34. doi: 10.1097/QAD.0b013e32835c54d8. PMID 23169332
- [Result] Jain V, Liegler T, Kabami J, Chamie G, Clark TD, Black D, Geng EH, Kwarisiima D, Wong JK, Abdel-Mohsen M, Sonawane N, Aweeka FT, Thirumurthy H, Petersen ML, Charlebois ED, Kamya MR, Havlir DV; SEARCH Collaboration. Assessment of population-based HIV RNA levels in a rural east African setting using a fingerprick-based blood collection method. Clin Infect Dis. 2013 Feb;56(4):598-605. doi: 10.1093/cid/cis881. Epub 2012 Dec 12. PMID 23243180
- [Result] Namusobya J, Semitala FC, Amanyire G, Kabami J, Chamie G, Bogere J, Jain V, Clark TD, Charlebois E, Havlir DV, Kamya M, Geng EH. High retention in care among HIV-infected patients entering care with CD4 levels >350 cells/muL under routine program conditions in Uganda. Clin Infect Dis. 2013 Nov;57(9):1343-50. doi: 10.1093/cid/cit490. Epub 2013 Jul 29. PMID 23899683
- [Result] Jain V, Byonanebye DM, Liegler T, Kwarisiima D, Chamie G, Kabami J, Petersen ML, Balzer LB, Clark TD, Black D, Thirumurthy H, Geng EH, Charlebois ED, Amanyire G, Kamya MR, Havlir DV; SEARCH Collaboration. Changes in population HIV RNA levels in Mbarara, Uganda, during scale-up of HIV antiretroviral therapy access. J Acquir Immune Defic Syndr. 2014 Mar 1;65(3):327-32. doi: 10.1097/QAI.0000000000000021. PMID 24146022
- [Result] Chamie G, Kwarisiima D, Clark TD, Kabami J, Jain V, Geng E, Balzer LB, Petersen ML, Thirumurthy H, Charlebois ED, Kamya MR, Havlir DV. Uptake of community-based HIV testing during a multi-disease health campaign in rural Uganda. PLoS One. 2014 Jan 2;9(1):e84317. doi: 10.1371/journal.pone.0084317. eCollection 2014. PMID 24392124
- [Result] Kotwani P, Kwarisiima D, Clark TD, Kabami J, Geng EH, Jain V, Chamie G, Petersen ML, Thirumurthy H, Kamya MR, Charlebois ED, Havlir DV; SEARCH Collaboration. Epidemiology and awareness of hypertension in a rural Ugandan community: a cross-sectional study. BMC Public Health. 2013 Dec 9;13:1151. doi: 10.1186/1471-2458-13-1151. PMID 24321133
- [Result] Kotwani P, Balzer L, Kwarisiima D, Clark TD, Kabami J, Byonanebye D, Bainomujuni B, Black D, Chamie G, Jain V, Thirumurthy H, Kamya MR, Geng EH, Petersen ML, Havlir DV, Charlebois ED; SEARCH Collaboration. Evaluating linkage to care for hypertension after community-based screening in rural Uganda. Trop Med Int Health. 2014 Apr;19(4):459-68. doi: 10.1111/tmi.12273. Epub 2014 Feb 3. PMID 24495307
- [Result] Jain V, Byonanebye DM, Amanyire G, Kwarisiima D, Black D, Kabami J, Chamie G, Clark TD, Rooney JF, Charlebois ED, Kamya MR, Havlir DV; SEARCH Collaboration. Successful antiretroviral therapy delivery and retention in care among asymptomatic individuals with high CD4+ T-cell counts above 350 cells/mul in rural Uganda. AIDS. 2014 Sep 24;28(15):2241-9. doi: 10.1097/QAD.0000000000000401. PMID 25022596
- [Result] Kwarisiima D, Balzer L, Heller D, Kotwani P, Chamie G, Clark T, Ayieko J, Mwangwa F, Jain V, Byonanebye D, Petersen M, Havlir D, Kamya MR. Population-Based Assessment of Hypertension Epidemiology and Risk Factors among HIV-Positive and General Populations in Rural Uganda. PLoS One. 2016 May 27;11(5):e0156309. doi: 10.1371/journal.pone.0156309. eCollection 2016. PMID 27232186
- [Result] Chamie G, Clark TD, Kabami J, Kadede K, Ssemmondo E, Steinfeld R, Lavoy G, Kwarisiima D, Sang N, Jain V, Thirumurthy H, Liegler T, Balzer LB, Petersen ML, Cohen CR, Bukusi EA, Kamya MR, Havlir DV, Charlebois ED. A hybrid mobile approach for population-wide HIV testing in rural east Africa: an observational study. Lancet HIV. 2016 Mar;3(3):e111-9. doi: 10.1016/S2352-3018(15)00251-9. Epub 2016 Jan 26. PMID 26939734
- [Result] Katrak S, Day N, Ssemmondo E, Kwarisiima D, Midekisa A, Greenhouse B, Kamya M, Havlir D, Dorsey G. Community-wide Prevalence of Malaria Parasitemia in HIV-Infected and Uninfected Populations in a High-Transmission Setting in Uganda. J Infect Dis. 2016 Jun 15;213(12):1971-8. doi: 10.1093/infdis/jiw057. Epub 2016 Feb 10. PMID 26908725
- [Result] Kadede K, Ruel T, Kabami J, Ssemmondo E, Sang N, Kwarisiima D, Bukusi E, Cohen CR, Liegler T, Clark TD, Charlebois ED, Petersen ML, Kamya MR, Havlir DV, Chamie G; SEARCH team. Increased adolescent HIV testing with a hybrid mobile strategy in Uganda and Kenya. AIDS. 2016 Sep 10;30(14):2121-6. doi: 10.1097/QAD.0000000000001180. PMID 27258399
- [Result] Jain V, Chang W, Byonanebye DM, Owaraganise A, Twinomuhwezi E, Amanyire G, Black D, Marseille E, Kamya MR, Havlir DV, Kahn JG. Estimated Costs for Delivery of HIV Antiretroviral Therapy to Individuals with CD4+ T-Cell Counts >350 cells/uL in Rural Uganda. PLoS One. 2015 Dec 3;10(12):e0143433. doi: 10.1371/journal.pone.0143433. eCollection 2015. PMID 26632823
- [Result] Balzer LB, Petersen ML, van der Laan MJ; SEARCH Collaboration. Targeted estimation and inference for the sample average treatment effect in trials with and without pair-matching. Stat Med. 2016 Sep 20;35(21):3717-32. doi: 10.1002/sim.6965. Epub 2016 Apr 18. PMID 27087478
- [Result] Thirumurthy H, Jakubowski A, Camlin C, Kabami J, Ssemmondo E, Elly A, Mwai D, Clark T, Cohen C, Bukusi E, Kamya M, Petersen M, Havlir D, Charlebois ED. Expectations about future health and longevity in Kenyan and Ugandan communities receiving a universal test-and-treat intervention in the SEARCH trial. AIDS Care. 2016;28 Suppl 3(Suppl 3):90-8. doi: 10.1080/09540121.2016.1178959. PMID 27421056
- [Result] Maeri I, El Ayadi A, Getahun M, Charlebois E, Akatukwasa C, Tumwebaze D, Itiakorit H, Owino L, Kwarisiima D, Ssemmondo E, Sang N, Kabami J, Clark TD, Petersen M, Cohen CR, Bukusi EA, Kamya M, Havlir D, Camlin CS; SEARCH Collaboration. "How can I tell?" Consequences of HIV status disclosure among couples in eastern African communities in the context of an ongoing HIV "test-and-treat" trial. AIDS Care. 2016;28 Suppl 3(Suppl 3):59-66. doi: 10.1080/09540121.2016.1168917. PMID 27421052
- [Result] Camlin CS, Ssemmondo E, Chamie G, El Ayadi AM, Kwarisiima D, Sang N, Kabami J, Charlebois E, Petersen M, Clark TD, Bukusi EA, Cohen CR, R Kamya M, Havlir D; SEARCH Collaboration. Men "missing" from population-based HIV testing: insights from qualitative research. AIDS Care. 2016;28 Suppl 3(Suppl 3):67-73. doi: 10.1080/09540121.2016.1164806. PMID 27421053
- [Result] Jain V, Petersen ML, Liegler T, Byonanebye DM, Kwarisiima D, Chamie G, Sang N, Black D, Clark TD, Ladai A, Plenty A, Kabami J, Ssemmondo E, Bukusi EA, Cohen CR, Charlebois ED, Kamya MR, Havlir DV; SEARCH Collaboration. Population levels and geographical distribution of HIV RNA in rural Ugandan and Kenyan communities, including serodiscordant couples: a cross-sectional analysis. Lancet HIV. 2017 Mar;4(3):e122-e133. doi: 10.1016/S2352-3018(16)30220-X. Epub 2016 Dec 16. PMID 27989576
- [Result] Brown LB, Havlir DV, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Jain V, Ruel T, Clark T, Chamie G, Bukusi EA, Cohen CR, Kamya MR, Petersen ML, Charlebois ED; SEARCH Collaboration. High levels of retention in care with streamlined care and universal test and treat in East Africa. AIDS. 2016 Nov 28;30(18):2855-2864. doi: 10.1097/QAD.0000000000001250. PMID 27603290
- [Result] Chang W, Chamie G, Mwai D, Clark TD, Thirumurthy H, Charlebois ED, Petersen M, Kabami J, Ssemmondo E, Kadede K, Kwarisiima D, Sang N, Bukusi EA, Cohen CR, Kamya M, Havlir DV, Kahn JG. Implementation and Operational Research: Cost and Efficiency of a Hybrid Mobile Multidisease Testing Approach With High HIV Testing Coverage in East Africa. J Acquir Immune Defic Syndr. 2016 Nov 1;73(3):e39-e45. doi: 10.1097/QAI.0000000000001141. PMID 27741031
- [Result] Brown LB, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Jain V, Ruel T, Clark T, Black D, Chamie G, Bukusi EA, Cohen CR, Kamya MR, Petersen ML, Charlebois ED, Havlir DV. Predictors of Retention in HIV Care Among Youth (15-24) in a Universal Test-and-Treat Setting in Rural Kenya. J Acquir Immune Defic Syndr. 2017 Sep 1;76(1):e15-e18. doi: 10.1097/QAI.0000000000001390. No abstract available. PMID 28394821
- [Result] Ssemmondo E, Mwangwa F, Kironde JL, Kwarisiima D, Clark TD, Marquez C, Charlebois ED, Petersen ML, Kamya MR, Havlir DV, Chamie G; SEARCH Collaboration. Implementation and Operational Research: Population-Based Active Tuberculosis Case Finding During Large-Scale Mobile HIV Testing Campaigns in Rural Uganda. J Acquir Immune Defic Syndr. 2016 Nov 1;73(3):e46-e50. doi: 10.1097/QAI.0000000000001142. PMID 27741032
- [Result] Petersen M, Balzer L, Kwarsiima D, Sang N, Chamie G, Ayieko J, Kabami J, Owaraganise A, Liegler T, Mwangwa F, Kadede K, Jain V, Plenty A, Brown L, Lavoy G, Schwab J, Black D, van der Laan M, Bukusi EA, Cohen CR, Clark TD, Charlebois E, Kamya M, Havlir D. Association of Implementation of a Universal Testing and Treatment Intervention With HIV Diagnosis, Receipt of Antiretroviral Therapy, and Viral Suppression in East Africa. JAMA. 2017 Jun 6;317(21):2196-2206. doi: 10.1001/jama.2017.5705. PMID 28586888
- [Result] Zheng W, Balzer L, van der Laan M, Petersen M; SEARCH Collaboration. Constrained binary classification using ensemble learning: an application to cost-efficient targeted PrEP strategies. Stat Med. 2018 Jan 30;37(2):261-279. doi: 10.1002/sim.7296. Epub 2017 Apr 6. PMID 28384841
- [Result] Mwangwa F, Chamie G, Kwarisiima D, Ayieko J, Owaraganise A, Ruel TD, Plenty A, Tram KH, Clark TD, Cohen CR, Bukusi EA, Petersen M, Kamya MR, Charlebois ED, Havlir DV, Marquez C. Gaps in the Child Tuberculosis Care Cascade in 32 Rural Communities in Uganda and Kenya. J Clin Tuberc Other Mycobact Dis. 2017 Dec;9:24-29. doi: 10.1016/j.jctube.2017.10.003. PMID 29291251
- [Result] Camlin CS, Charlebois ED, Geng E, Semitala F, Wallenta J, Getahun M, Kampiire L, Bukusi EA, Sang N, Kwarisiima D, Clark TD, Petersen ML, Kamya MR, Havlir DV. Redemption of the "spoiled identity:" the role of HIV-positive individuals in HIV care cascade interventions. J Int AIDS Soc. 2017 Dec;20(4):e25023. doi: 10.1002/jia2.25023. PMID 29210185
- [Result] Koss CA, Ayieko J, Mwangwa F, Owaraganise A, Kwarisiima D, Balzer LB, Plenty A, Sang N, Kabami J, Ruel TD, Black D, Camlin CS, Cohen CR, Bukusi EA, Clark TD, Charlebois ED, Petersen ML, Kamya MR, Havlir DV; SEARCH Collaboration. Early Adopters of Human Immunodeficiency Virus Preexposure Prophylaxis in a Population-based Combination Prevention Study in Rural Kenya and Uganda. Clin Infect Dis. 2018 Nov 28;67(12):1853-1860. doi: 10.1093/cid/ciy390. PMID 29741594
- [Result] Camlin CS, Koss CA, Getahun M, Owino L, Itiakorit H, Akatukwasa C, Maeri I, Bakanoma R, Onyango A, Atwine F, Ayieko J, Kabami J, Mwangwa F, Atukunda M, Owaraganise A, Kwarisiima D, Sang N, Bukusi EA, Kamya MR, Petersen ML, Cohen CR, Charlebois ED, Havlir DV. Understanding Demand for PrEP and Early Experiences of PrEP Use Among Young Adults in Rural Kenya and Uganda: A Qualitative Study. AIDS Behav. 2020 Jul;24(7):2149-2162. doi: 10.1007/s10461-020-02780-x. PMID 31955361
- [Result] Heller DJ, Balzer LB, Kazi D, Charlebois ED, Kwarisiima D, Mwangwa F, Jain V, Kotwani P, Chamie G, Cohen CR, Clark TD, Ayieko J, Byonanabye DM, Petersen M, Kamya MR, Havlir D, Kahn JG. Hypertension testing and treatment in Uganda and Kenya through the SEARCH study: An implementation fidelity and outcome evaluation. PLoS One. 2020 Jan 15;15(1):e0222801. doi: 10.1371/journal.pone.0222801. eCollection 2020. PMID 31940346
- [Result] Brown LB, Balzer LB, Kabami J, Kwarisiima D, Sang N, Ayieko J, Chen Y, Chamie G, Charlebois ED, Camlin CS, Cohen CR, Bukusi E, Kamya MR, Moody J, Havlir DV, Petersen ML. The Influence of Social Networks on Antiretroviral Therapy Initiation Among HIV-Infected Antiretroviral Therapy-Naive Youth in Rural Kenya and Uganda. J Acquir Immune Defic Syndr. 2020 Jan 1;83(1):9-15. doi: 10.1097/QAI.0000000000002199. PMID 31809357
- [Result] Olilo WA, Petersen ML, Koss CA, Wafula E, Kwarisiima D, Kadede K, Clark TD, Cohen CR, Bukusi EA, Kamya MR, Charlebois ED, Havlir DV, Ayieko J; SEARCH Collaboration. Pre-exposure Prophylaxis (PrEP) Uptake Among Older Individuals in Rural Western Kenya. J Acquir Immune Defic Syndr. 2019 Dec 1;82(4):e50-e53. doi: 10.1097/QAI.0000000000002150. No abstract available. PMID 31490343
- [Result] Chamie G, Kamya MR, Petersen ML, Havlir DV. Reaching 90-90-90 in rural communities in East Africa: lessons from the Sustainable East Africa Research in Community Health Trial. Curr Opin HIV AIDS. 2019 Nov;14(6):449-454. doi: 10.1097/COH.0000000000000585. PMID 31589172
- [Result] Havlir DV, Balzer LB, Charlebois ED, Clark TD, Kwarisiima D, Ayieko J, Kabami J, Sang N, Liegler T, Chamie G, Camlin CS, Jain V, Kadede K, Atukunda M, Ruel T, Shade SB, Ssemmondo E, Byonanebye DM, Mwangwa F, Owaraganise A, Olilo W, Black D, Snyman K, Burger R, Getahun M, Achando J, Awuonda B, Nakato H, Kironde J, Okiror S, Thirumurthy H, Koss C, Brown L, Marquez C, Schwab J, Lavoy G, Plenty A, Mugoma Wafula E, Omanya P, Chen YH, Rooney JF, Bacon M, van der Laan M, Cohen CR, Bukusi E, Kamya MR, Petersen M. HIV Testing and Treatment with the Use of a Community Health Approach in Rural Africa. N Engl J Med. 2019 Jul 18;381(3):219-229. doi: 10.1056/NEJMoa1809866. PMID 31314966
- [Result] Tram KH, Mwangwa F, Chamie G, Atukunda M, Owaraganise A, Ayieko J, Jain V, Clark TD, Kwarisiima D, Petersen ML, Kamya MR, Charlebois ED, Havlir DV, Marquez C; SEARCH collaboration. Predictors of isoniazid preventive therapy completion among HIV-infected patients receiving differentiated and non-differentiated HIV care in rural Uganda. AIDS Care. 2020 Jan;32(1):119-127. doi: 10.1080/09540121.2019.1619661. Epub 2019 Jun 10. PMID 31181961
- [Result] Kwarisiima D, Atukunda M, Owaraganise A, Chamie G, Clark T, Kabami J, Jain V, Byonanebye D, Mwangwa F, Balzer LB, Charlebois E, Kamya MR, Petersen M, Havlir DV, Brown LB. Hypertension control in integrated HIV and chronic disease clinics in Uganda in the SEARCH study. BMC Public Health. 2019 May 6;19(1):511. doi: 10.1186/s12889-019-6838-6. PMID 31060545
- [Result] Mayer CM, Owaraganise A, Kabami J, Kwarisiima D, Koss CA, Charlebois ED, Kamya MR, Petersen ML, Havlir DV, Jewell BL. Distance to clinic is a barrier to PrEP uptake and visit attendance in a community in rural Uganda. J Int AIDS Soc. 2019 Apr;22(4):e25276. doi: 10.1002/jia2.25276. PMID 31037845
- [Result] Camlin CS, Akullian A, Neilands TB, Getahun M, Bershteyn A, Ssali S, Geng E, Gandhi M, Cohen CR, Maeri I, Eyul P, Petersen ML, Havlir DV, Kamya MR, Bukusi EA, Charlebois ED. Gendered dimensions of population mobility associated with HIV across three epidemics in rural Eastern Africa. Health Place. 2019 May;57:339-351. doi: 10.1016/j.healthplace.2019.05.002. Epub 2019 May 29. PMID 31152972
- [Result] Ayieko J, Petersen ML, Charlebois ED, Brown LB, Clark TD, Kwarisiima D, Kamya MR, Cohen CR, Bukusi EA, Havlir DV, Van Rie A. A Patient-Centered Multicomponent Strategy for Accelerated Linkage to Care Following Community-Wide HIV Testing in Rural Uganda and Kenya. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):414-422. doi: 10.1097/QAI.0000000000001939. PMID 30807481
- [Result] Brown LB, Getahun M, Ayieko J, Kwarisiima D, Owaraganise A, Atukunda M, Olilo W, Clark T, Bukusi EA, Cohen CR, Kamya MR, Petersen ML, Charlebois ED, Havlir DV, Camlin CS. Factors predictive of successful retention in care among HIV-infected men in a universal test-and-treat setting in Uganda and Kenya: A mixed methods analysis. PLoS One. 2019 Jan 23;14(1):e0210126. doi: 10.1371/journal.pone.0210126. eCollection 2019. PMID 30673744
- [Result] Shade SB, Osmand T, Luo A, Aine R, Assurah E, Mwebaza B, Mwai D, Owaraganise A, Mwangwa F, Ayieko J, Black D, Brown LB, Clark TD, Kwarisiima D, Thirumurthy H, Cohen CR, Bukusi EA, Charlebois ED, Balzer L, Kamya MR, Petersen ML, Havlir DV, Jain V. Costs of streamlined HIV care delivery in rural Ugandan and Kenyan clinics in the SEARCH Studys. AIDS. 2018 Sep 24;32(15):2179-2188. doi: 10.1097/QAD.0000000000001958. PMID 30134294
- [Result] Marquez C, Atukunda M, Balzer LB, Chamie G, Kironde J, Ssemmondo E, Ruel TD, Mwangwa F, Tram KH, Clark TD, Kwarisiima D, Petersen M, Kamya MR, Charlebois ED, Havlir DV. The age-specific burden and household and school-based predictors of child and adolescent tuberculosis infection in rural Uganda. PLoS One. 2020 Jan 29;15(1):e0228102. doi: 10.1371/journal.pone.0228102. eCollection 2020. PMID 31995631
- [Result] Havlir D, Lockman S, Ayles H, Larmarange J, Chamie G, Gaolathe T, Iwuji C, Fidler S, Kamya M, Floyd S, Moore J, Hayes R, Petersen M, Dabis F; (Universal Test, Treat Trials) UT3 Consortium. What do the Universal Test and Treat trials tell us about the path to HIV epidemic control? J Int AIDS Soc. 2020 Feb;23(2):e25455. doi: 10.1002/jia2.25455. PMID 32091179
- [Result] Muiru AN, Charlebois ED, Balzer LB, Kwarisiima D, Elly A, Black D, Okiror S, Kabami J, Atukunda M, Snyman K, Petersen M, Kamya M, Havlir D, Estrella MM, Hsu CY. The epidemiology of chronic kidney disease (CKD) in rural East Africa: A population-based study. PLoS One. 2020 Mar 4;15(3):e0229649. doi: 10.1371/journal.pone.0229649. eCollection 2020. PMID 32130245
- [Result] Koss CA, Charlebois ED, Ayieko J, Kwarisiima D, Kabami J, Balzer LB, Atukunda M, Mwangwa F, Peng J, Mwinike Y, Owaraganise A, Chamie G, Jain V, Sang N, Olilo W, Brown LB, Marquez C, Zhang K, Ruel TD, Camlin CS, Rooney JF, Black D, Clark TD, Gandhi M, Cohen CR, Bukusi EA, Petersen ML, Kamya MR, Havlir DV; SEARCH Collaboration. Uptake, engagement, and adherence to pre-exposure prophylaxis offered after population HIV testing in rural Kenya and Uganda: 72-week interim analysis of observational data from the SEARCH study. Lancet HIV. 2020 Apr;7(4):e249-e261. doi: 10.1016/S2352-3018(19)30433-3. Epub 2020 Feb 19. PMID 32087152
- [Result] Chamie G, Hickey MD, Kwarisiima D, Ayieko J, Kamya MR, Havlir DV. Universal HIV Testing and Treatment (UTT) Integrated with Chronic Disease Screening and Treatment: the SEARCH study. Curr HIV/AIDS Rep. 2020 Aug;17(4):315-323. doi: 10.1007/s11904-020-00500-7. PMID 32507985
- [Result] Kabami J, Balzer LB, Saddiki H, Ayieko J, Kwarisiima D, Atukunda M, Charlebois ED, Clark TD, Koss CA, Ruel T, Bukusi EA, Cohen CR, Musoke P, Petersen ML, Havlir DV, Kamya MR, Chamie G. Population-level viral suppression among pregnant and postpartum women in a universal test and treat trial. AIDS. 2020 Jul 15;34(9):1407-1415. doi: 10.1097/QAD.0000000000002564. PMID 32472768
- [Result] Hickey MD, Ayieko J, Kwarisiima D, Opel FJ, Owaraganise A, Balzer LB, Chamie G, Jain V, Peng J, Camlin C, Charlebois ED, Cohen CR, Bukusi EA, Kamya MR, Petersen ML, Havlir DV. Improved Viral Suppression With Streamlined Care in the SEARCH Study. J Acquir Immune Defic Syndr. 2020 Dec 15;85(5):571-578. doi: 10.1097/QAI.0000000000002508. PMID 32991337
- [Result] Camlin CS, Charlebois ED, Getahun M, Akatukwasa C, Atwine F, Itiakorit H, Bakanoma R, Maeri I, Owino L, Onyango A, Chamie G, Clark TD, Cohen CR, Kwarisiima D, Kabami J, Sang N, Kamya MR, Bukusi EA, Petersen ML, V Havlir D. Pathways for reduction of HIV-related stigma: a model derived from longitudinal qualitative research in Kenya and Uganda. J Int AIDS Soc. 2020 Dec;23(12):e25647. doi: 10.1002/jia2.25647. PMID 33283986
- [Result] Koss CA, Havlir DV, Ayieko J, Kwarisiima D, Kabami J, Chamie G, Atukunda M, Mwinike Y, Mwangwa F, Owaraganise A, Peng J, Olilo W, Snyman K, Awuonda B, Clark TD, Black D, Nugent J, Brown LB, Marquez C, Okochi H, Zhang K, Camlin CS, Jain V, Gandhi M, Cohen CR, Bukusi EA, Charlebois ED, Petersen ML, Kamya MR, Balzer LB. HIV incidence after pre-exposure prophylaxis initiation among women and men at elevated HIV risk: A population-based study in rural Kenya and Uganda. PLoS Med. 2021 Feb 9;18(2):e1003492. doi: 10.1371/journal.pmed.1003492. eCollection 2021 Feb. PMID 33561143
- [Result] Nyabuti MN, Petersen ML, Bukusi EA, Kamya MR, Mwangwa F, Kabami J, Sang N, Charlebois ED, Balzer LB, Schwab JD, Camlin CS, Black D, Clark TD, Chamie G, Havlir DV, Ayieko J. Characteristics of HIV seroconverters in the setting of universal test and treat: Results from the SEARCH trial in rural Uganda and Kenya. PLoS One. 2021 Feb 5;16(2):e0243167. doi: 10.1371/journal.pone.0243167. eCollection 2021. PMID 33544717
- [Result] Shade SB, Osmand T, Kwarisiima D, Brown LB, Luo A, Mwebaza B, Mwesigye AR, Kwizera E, Imukeka H, Mwanga F, Ayieko J, Owaraganise A, Bukusi EA, Cohen CR, Charlebois ED, Black D, Clark TD, Petersen ML, Kamya MR, Havlir DV, Jain V. Costs of integrating hypertension care into HIV care in rural East African clinics. AIDS. 2021 May 1;35(6):911-919. doi: 10.1097/QAD.0000000000002834. PMID 33821821
- [Result] Chamie G, Kwarisiima D, Ndyabakira A, Marson K, Camlin CS, Havlir DV, Kamya MR, Thirumurthy H. Financial incentives and deposit contracts to promote HIV retesting in Uganda: A randomized trial. PLoS Med. 2021 May 4;18(5):e1003630. doi: 10.1371/journal.pmed.1003630. eCollection 2021 May. PMID 33945526
- [Derived] Camlin CS, Gutin SA, Charlebois ED, Neilands TB, Balzer LB, Petersen ML, Chamie G, Cohen CR, Bukusi EA, Kamya MR, Havlir DV, Ayieko J. Metrics of Mobility by Sex are Associated with HIV Incidence in Rural Kenya and Uganda. AIDS Behav. 2025 Sep;29(9):2869-2881. doi: 10.1007/s10461-025-04743-6. Epub 2025 May 6. PMID 40327268
- [Derived] Abbott R, Landsiedel K, Atukunda M, Puryear SB, Chamie G, Hahn JA, Mwangwa F, Kakande E, Petersen ML, Havlir DV, Charlebois E, Balzer LB, Kamya MR, Marquez C. Incident Tuberculosis Infection Is Associated With Alcohol Use in Adults in Rural Uganda. Clin Infect Dis. 2025 Mar 17;80(3):562-565. doi: 10.1093/cid/ciae304. PMID 38824440
- [Derived] Marquez C, Atukunda M, Nugent J, Charlebois ED, Chamie G, Mwangwa F, Ssemmondo E, Kironde J, Kabami J, Owaraganise A, Kakande E, Ssekaynzi B, Abbott R, Ayieko J, Ruel T, Kwariisima D, Kamya M, Petersen M, Havlir DV, Balzer LB. Community-Wide Universal HIV Test and Treat Intervention Reduces Tuberculosis Transmission in Rural Uganda: A Cluster-Randomized Trial. Clin Infect Dis. 2024 Jun 14;78(6):1601-1607. doi: 10.1093/cid/ciad776. PMID 38226445
- [Derived] Ayieko J, Charlebois ED, Maeri I, Owino L, Thorp M, Bukusi EA, Petersen ML, Kamya MR, Havlir DV, Camlin CS. Improving care engagement for mobile people living with HIV in rural western Kenya. PLoS One. 2023 Nov 22;18(11):e0288087. doi: 10.1371/journal.pone.0288087. eCollection 2023. PMID 37992063
- [Derived] Puryear SB, Ayieko J, Hahn JA, Mucunguzi A, Owaraganise A, Schwab J, Balzer LB, Kwarisiima D, Charlebois ED, Cohen CR, Bukusi EA, Petersen ML, Havlir DV, Kamya MR, Chamie G. Universal HIV Testing and Treatment With Patient-Centered Care Improves ART Uptake and Viral Suppression Among Adults Reporting Hazardous Alcohol Use in Uganda and Kenya. J Acquir Immune Defic Syndr. 2023 Sep 1;94(1):37-45. doi: 10.1097/QAI.0000000000003226. PMID 37220015
- [Derived] Maeri I, Eyul P, Getahun M, Hatchett K, Owino L, Akatukwasa C, Itiakorit H, Gutin SA, Johnson-Peretz J, Ssali S, Cohen CR, Bukusi EA, Kamya MR, Charlebois ED, Camlin CS. Nothing about us without us: Community-based participatory research to improve HIV care for mobile patients in Kenya and Uganda. Soc Sci Med. 2023 Feb;318:115471. doi: 10.1016/j.socscimed.2022.115471. Epub 2022 Oct 28. PMID 36628879
- [Derived] Camlin CS, Getahun M, Koss CA, Owino L, Akatukwasa C, Itiakorit H, Onyango A, Bakanoma R, Atwine F, Maeri I, Ayieko J, Atukunda M, Owaraganise A, Mwangwa F, Sang N, Kabami J, Kaplan RL, Chamie G, Petersen ML, Cohen CR, Bukusi EA, Kamya MR, Havlir DV, Charlebois ED. Providers' Attitudes and Experiences with Pre-Exposure Prophylaxis Implementation in a Population-Based Study in Kenya and Uganda. AIDS Patient Care STDS. 2022 Oct;36(10):396-404. doi: 10.1089/apc.2022.0084. Epub 2022 Oct 5. PMID 36201226
- [Derived] Jakubowski A, Kabami J, Balzer LB, Ayieko J, Charlebois ED, Owaraganise A, Marquez C, Clark TD, Black D, Shade SB, Chamie G, Cohen CR, Bukusi EA, Kamya MR, Petersen M, Havlir DV, Thirumurthy H. Effect of universal HIV testing and treatment on socioeconomic wellbeing in rural Kenya and Uganda: a cluster-randomised controlled trial. Lancet Glob Health. 2022 Jan;10(1):e96-e104. doi: 10.1016/S2214-109X(21)00458-7. PMID 34919862
- [Derived] Mwangwa F, Getahun M, Itiakorit H, Jain V, Ayieko J, Owino L, Akatukwasa C, Maeri I, Koss CA, Chamie G, Clark TD, Kabami J, Atukunda M, Kwarisiima D, Sang N, Bukusi EA, Kamya MR, Petersen ML, Cohen CR, Charlebois ED, Havlir DV, Camlin CS. Provider and Patient Perspectives of Rapid ART Initiation and Streamlined HIV Care: Qualitative Insights From Eastern African Communities. J Int Assoc Provid AIDS Care. 2021 Jan-Dec;20:23259582211053518. doi: 10.1177/23259582211053518. PMID 34841945
- [Derived] Hickey MD, Ayieko J, Owaraganise A, Sim N, Balzer LB, Kabami J, Atukunda M, Opel FJ, Wafula E, Nyabuti M, Brown L, Chamie G, Jain V, Peng J, Kwarisiima D, Camlin CS, Charlebois ED, Cohen CR, Bukusi EA, Kamya MR, Petersen ML, Havlir DV. Effect of a patient-centered hypertension delivery strategy on all-cause mortality: Secondary analysis of SEARCH, a community-randomized trial in rural Kenya and Uganda. PLoS Med. 2021 Sep 20;18(9):e1003803. doi: 10.1371/journal.pmed.1003803. eCollection 2021 Sep. PMID 34543267
- [Derived] Ayieko J, Petersen ML, Kabami J, Mwangwa F, Opel F, Nyabuti M, Charlebois ED, Peng J, Koss CA, Balzer LB, Chamie G, Bukusi EA, Kamya MR, Havlir DV. Uptake and outcomes of a novel community-based HIV post-exposure prophylaxis (PEP) programme in rural Kenya and Uganda. J Int AIDS Soc. 2021 Jun;24(6):e25670. doi: 10.1002/jia2.25670. PMID 34152067
- [Derived] Kamya MR, Petersen ML, Kabami J, Ayieko J, Kwariisima D, Sang N, Clark TD, Schwab J, Charlebois ED, Cohen CR, Bukusi EA, Peng J, Jain V, Chen YH, Chamie G, Balzer LB, Havlir DV. SEARCH Human Immunodeficiency Virus (HIV) Streamlined Treatment Intervention Reduces Mortality at a Population Level in Men With Low CD4 Counts. Clin Infect Dis. 2021 Oct 5;73(7):e1938-e1945. doi: 10.1093/cid/ciaa1782. PMID 33783495
- [Derived] Ayieko J, Brown L, Anthierens S, Van Rie A, Getahun M, Charlebois ED, Petersen ML, Clark TD, Kamya MR, Cohen CR, Bukusi EA, Havlir DV, Camlin CS. "Hurdles on the path to 90-90-90 and beyond": Qualitative analysis of barriers to engagement in HIV care among individuals in rural East Africa in the context of test-and-treat. PLoS One. 2018 Aug 30;13(8):e0202990. doi: 10.1371/journal.pone.0202990. eCollection 2018. PMID 30161172
- [Derived] Camlin CS, Akullian A, Neilands TB, Getahun M, Eyul P, Maeri I, Ssali S, Geng E, Gandhi M, Cohen CR, Kamya MR, Odeny T, Bukusi EA, Charlebois ED. Population mobility associated with higher risk sexual behaviour in eastern African communities participating in a Universal Testing and Treatment trial. J Int AIDS Soc. 2018 Jul;21 Suppl 4(Suppl Suppl 4):e25115. doi: 10.1002/jia2.25115. PMID 30027668
- [Derived] Jakubowski A, Snyman K, Kwarisiima D, Sang N, Burger R, Balzer L, Clark T, Chamie G, Shade S, Cohen C, Bukusi E, Charlebois E, Kamya M, Petersen M, Havlir D, Thirumurthy H. High CD4 counts associated with better economic outcomes for HIV-positive adults and their HIV-negative household members in the SEARCH Trial. PLoS One. 2018 Jun 26;13(6):e0198912. doi: 10.1371/journal.pone.0198912. eCollection 2018. PMID 29944678
- [Derived] Kwarisiima D, Kamya MR, Owaraganise A, Mwangwa F, Byonanebye DM, Ayieko J, Plenty A, Black D, Clark TD, Nzarubara B, Snyman K, Brown L, Bukusi E, Cohen CR, Geng EH, Charlebois ED, Ruel TD, Petersen ML, Havlir D, Jain V. High rates of viral suppression in adults and children with high CD4+ counts using a streamlined ART delivery model in the SEARCH trial in rural Uganda and Kenya. J Int AIDS Soc. 2017 Jul 21;20(Suppl 4):21673. doi: 10.7448/IAS.20.5.21673. PMID 28770596
- See also: SEARCH Collaboration website — http://www.searchendaids.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 communities were enrolled and randomized to the intervention and control (16 per arm in each stage). We enrolled 150,395 community residents aged 15+ years at study baseline in Stage 1. At the start of Stage 2, 184,091 community residents (including in-migrants) aged 15+ years were enrolled. The analytic population for each endpoint is detailed in the Outcomes section.
Units Other Than Participants: Communites
Groups:
- Intervention: Intervention arm first stage: annual universal community-based HIV and multi-disease testing; ART for all HIV+; ART delivery using streamlined patient-centered care
  Intervention arm second stage: Baseline universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care; targeted population-level PrEP
- Control: Active Comparator arm first stage: Baseline universal community-based HIV and multi-disease testing; ART eligibility and delivery by country standard of care
  Active Comparator arm second stage
Period: Stage 1
Arm/Group | Intervention | Control
Started | 79818; 16 Communites (Describes # of participants who were residents and aged 15+yrs at baseline) | 70577; 16 Communites (Describes # of participants who were residents and aged 15+yrs at baseline)
Completed | 71028; 16 Communites | 62912; 16 Communites
Not Completed | 8790; 0 Communites | 7665; 0 Communites
Period: Stage 2
Arm/Group | Intervention | Control
Started | 91533; 16 Communites (Describes # of participants who were residents and aged 15+yrs at the start of Stage 2) | 92558; 16 Communites (Describes # of participants who were residents and aged 15+yrs at the start of Stage 2)
Completed | 5477; 16 Communites | 0; 0 Communites
Not Completed | 86056; 0 Communites | 92558; 16 Communites
Not completed — DSMB design modification | 86056 | 92558

BASELINE CHARACTERISTICS:
Population: Persons who were residents and aged 15+ years at baseline.
Groups:
- Intervention: Intervention arm first stage: Annual universal community- based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care
- Control: Active Comparator arm first stage: Baseline universal community-based HIV and multi-disease testing; ART eligibility and delivery by country standard of care
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 79818 | 70577 | 150395
Age, Customized [Count of Participants; unit: Participants]
  15-20 years | 20053 | 16602 | 36655
  21-49 years | 44047 | 39975 | 84022
  >=50 years | 15718 | 14000 | 29718
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43770 | 38644 | 82414
  Male | 36048 | 31933 | 67981
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 79818 | 70577 | 150395
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Marital Status [Count of Participants; unit: Participants] — Population: Marital status not reported by all participants
  Participants
    number analyzed (Participants) | 79604 | 70436 | 150040
    Single | 23692 | 19392 | 43084
    Married | 46684 | 42502 | 89186
    Widowed, divorced or separated | 9228 | 8542 | 17770
Marital status - polygamous marriage [Count of Participants; unit: Participants] — Population: Polygamous marriage status was not reported by all participants
  Participants
    number analyzed (Participants) | 79595 | 70429 | 150024
    (all) | 9575 | 9210 | 18785
Education [Count of Participants; unit: Participants] — Population: Education was not reported by all participants
  Participants
    number analyzed (Participants) | 79656 | 70404 | 150060
    Below primary school | 50912 | 45691 | 96603
    Completed primary school | 11478 | 10305 | 21783
    Any secondary school or higher | 17266 | 14408 | 31674
Occupation [Count of Participants; unit: Participants] — A formal sector occupation was defined as a teacher, student, government worker, military worker, health worker, or factory worker. A high-risk informal sector occupation was defined as a fishmonger, fisher, bar owner, bar worker, transportation worker, or tourism worker. A low-risk informal sector occupation was defined as a farmer, shopkeeper, market vendor, hotel worker, homemaker, household worker, construction worker, or miner. Population: Occupation not reported by all participants
  Participants
    number analyzed (Participants) | 79597 | 70434 | 150031
    Formal sector | 19753 | 15733 | 35486
    High-risk informal sector | 3235 | 4944 | 8179
    Low-risk informal sector | 48753 | 42341 | 91094
    Other | 3595 | 3201 | 6796
    No job or disabled | 4261 | 4215 | 8476
Household wealth index quintile [Count of Participants; unit: Participants] — Quintiles were based on a principle components analysis of the household wealth survey and were calculated at the level of the household. Population: Household wealth survey data was not collected on all households.
  Participants
    number analyzed (Participants) | 79619 | 70280 | 149899
    First, indicating least wealth | 12078 | 11876 | 23954
    Second | 13474 | 12652 | 26126
    Third | 15448 | 14371 | 29819
    Fourth | 17384 | 15703 | 33087
    Fifth, indicating most wealth | 21235 | 15678 | 36913
Stable residents [Count of Participants; unit: Participants] — Stable residents were defined as residents who had spent at least 6 months of the previous year in the trial community. Population: Two participants did not have data recorded to determine as stable resident.
  Participants
    number analyzed (Participants) | 79816 | 70577 | 150393
    (all) | 76111 | 67759 | 143870
Residents living with HIV [Count of Participants; unit: Participants] — Population: HIV status was not available for all participants
  Participants
    number analyzed (Participants) | 71605 | 63879 | 135484
    (all) | 7212 | 6317 | 13529
Residents with prevalent hypertension [Count of Participants; unit: Participants] — Previous or current self-report of prior diagnosis OR previous or current systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg on all 3 measurements at the health campaign or on all measures if < 3 measurements done Population: Adults 30 years of age or older were included in the analysis.
  Participants
    number analyzed (Participants) | 28877 | 26884 | 55761
    (all) | 5953 | 5911 | 11864

OUTCOME MEASURES:

1. Primary Outcome: Cumulative HIV Incidence
Description: Cumulative 3 year HIV incidence in men and women ages ≥15 years after the start of Phase I intervention.
  Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Baseline HIV- stable adult (15+years) residents
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Groups:
- Intervention: Annual universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care
- Control: Baseline community-based HIV and multi-disease testing; ART eligibility and delivery by country standard of care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 61676 | 55438
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 0.77 [0.60 to 0.93] | 0.81 [0.68 to 0.94]
Statistical Analysis 1: Comparison: Intervention vs Control; Comparison of Phase 1 arms; Test type: Other; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.77 to 1.17]

2. Primary Outcome: HIV Incidence
Description: HIV incidence rate in men and women ages ≥15 years after the start of Phase II intervention (started after 3 years of Phase I).
Time Frame: 3 years follow up
Population: Intervention population consists of persons aged 15+ years who initiated PrEP in Phase II intervention communities. The comparator population consists of propensity score matched historical controls from Phase I intervention communities. HIV testing was not comprehensively conducted during Phase 2.
Measure: Number (95% Confidence Interval); unit: Incident HIV per 100 person-year
Groups:
- Intervention: Baseline universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care; targeted population-level PrEP
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5477 | 2061
Incident HIV per 100 person-year | 0.35 [0.22 to 0.49] | 0.92 [0.49 to 1.41]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Other; Rate ratio = 0.26, 95% CI 2-sided [0.09 to 0.75]

3. Secondary Outcome: Incident TB Associated With HIV
Description: Cumulative incidence of TB or death due to illness among HIV+ population. Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Adults without active TB and with HIV at baseline
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7022 | 6148
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 3.7 [3.2 to 4.1] | 4.6 [4.1 to 5.2]

4. Secondary Outcome: Overall Mortality
Description: Mortality risk among HIV+ population. Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Known HIV+ at baseline
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 6971 | 6095
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 3.0 [2.6 to 3.4] | 3.9 [3.4 to 4.4]

5. Secondary Outcome: HIV-free Infant Survival
Description: Probability of an infant born to an HIV+ mother remaining alive and HIV uninfected.
  Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Infants born in study period to women with HIV
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 564 | 528
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 96.7 [94.4 to 99.0] | 93.6 [92.0 to 95.3]

6. Secondary Outcome: Percent of HIV+ Adults With HIV RNA <=500 c/mL
Description: Percent of HIV+ adults with HIV RNA <=500 c/mL. Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: HIV+ adults at year 3, including those out of care or without a prior HIV diagnosis
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 8399 | 7349
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 79 [77 to 81] | 68 [66 to 70]

7. Secondary Outcome: Time in Care for HIV+ Adults With Baseline Viremia
Description: Percent of time spent actively engaged in HIV care among HIV+ adults with baseline viremia
Time Frame: 3 years follow up
Population: HIV+ adults linked to care with baseline HIV RNA >=500 c/mL
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 330 | 238
percentage of days | 81 [79 to 83] | 73 [68 to 79]

8. Secondary Outcome: Cumulative Incidence of ART-initiation
Description: Proportion of baseline HIV+ ART-naive persons who initiate ART Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Baseline HIV+ without previous or current ART
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 3002 | 2950
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 83 [80 to 85] | 50 [46 to 54]

9. Secondary Outcome: Hypertension Control
Description: hypertension control (greater than or equal to 140 mg Hg systolic or 90 mg Hg diastolic after 3 repeated readings) at year 3 among adults aged >= 30 years with hypertension.
  Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: Hypertensive adults (aged 30+) at year 3
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11664 | 10935
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 47 [45 to 49] | 37 [35 to 40]

10. Secondary Outcome: Adherence to PrEP Treatment
Description: Number of patients with adherence to PrEP treatment (self reported adherence at >=1 visit)
Time Frame: 3 years follow up
Population: Persons who initiated PrEP eligible for a follow-up visit. No data were collected for the second stage in the control arm due to DSMB approved design modification.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 5398
Participants | 3282

11. Secondary Outcome: Average Adults' on- and Off-farm Employment
Description: HIV+ adults with on- and off-farm employment
Time Frame: 3 years follow up
Population: Subsample of baseline HIV+ working-age adults (18-65)
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Arm/Group | Intervention | Control
Number analyzed (Participants) | 1425 | 1443
cumulative events per 100 persons | 85.5 [83.1 to 88.0] | 82.4 [80 to 84.9]

12. Secondary Outcome: Year 3 Viremia Among ART-experienced Persons With Baseline Viremia
Description: Plasma HIV RNA <400 cps/ml Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 3 years follow up
Population: HIV+ ART experienced adults linked to care with baseline HIV RNA >=500 c/mL
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Arm/Group | Intervention | Control
Number analyzed (Participants) | 330 | 238
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 67 [59 to 74] | 47 [36 to 58]

13. Secondary Outcome: Linkage to Care
Description: Proportion of Persons Attending an HIV Clinic Visit by 30 Days After HIV Test Mean was calculated as the average across clusters of the cluster-level cumulative incidence.
Time Frame: 30 days after HIV test
Population: Persons testing HIV+ and not in care
Measure: Mean (95% Confidence Interval); unit: cumulative events per 100 persons
Units Other Than Participants: Communities
Groups:
- Intervention: Patient-centered Phone call
- Control: Standard of Care
Arm/Group | Intervention | Control
Number analyzed (Participants) | 68 | 62
Number analyzed (Communities) | 16 | 16
cumulative events per 100 persons | 41 [29 to 53] | 24 [13 to 35]

14. Secondary Outcome: HIV Incidence Rate
Description: HIV incidence rates during the first and third year of follow up; Results from the Control arm are not provided because annual HIV incidence was not measured in the control arm (annual HIV testing was only conducted in the intervention arm).
Time Frame: 3 years follow up
Population: HIV-negative adults in stage 1 intervention arm who had repeat HIV testing
Measure: Number (95% Confidence Interval); unit: per 100 person-years
Groups:
- Intervention Year 1: Third year of Stage 1 intervention
- Intervention Year 3: First year of Stage 1 Intervention: Annual universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care
Arm/Group | Intervention Year 1 | Intervention Year 3
Number analyzed (Participants) | 52474 | 58145
per 100 person-years | 0.43 [0.38 to 0.49] | 0.31 [0.26 to 0.36]

15. Secondary Outcome: Prevalence of Transmitted HIV Drug-resistance Mutations
Description: HIV NNRTI drug-resistance mutations found at baseline
Time Frame: Baseline
Population: ART naive HIV+ persons at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 74 | 107
Participants | 8 | 11

16. Secondary Outcome: Prevalence of Chronic Kidney Disease (CKD)
Description: Percentage of participants with chronic kidney disease (CKD)
Time Frame: 3 years follow up
Population: participants (age >=18) who had a home visit during follow up year 3
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2100 | 1505
Participants | 361 | 248

17. Secondary Outcome: Total Costs of Programming (ART)
Description: Cost of ART streamlined care delivery amount HIV+ persons
Time Frame: Follow up year 3
Population: Units are Intervention clinics using streamlined care; participants are HIV+ with at least one streamlined care visit
Measure: Mean (95% Confidence Interval); unit: USD per person year
Units Other Than Participants: Clinics
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7700 | 7700
Number analyzed (Clinics) | 17 | 17
USD per person year | 291 [279 to 303] | 221 [196 to 246]

ADVERSE EVENTS:
Time Frame: Phase I: 3 years Phase II: 3 years
Description: This was a community randomized community-based trial. In accordance with our approved data safety monitoring plan, adverse events were monitored and assessed in a different population of patients than all cause mortality. Adverse events were only monitored for participants who received any biomedical treatment or prevention intervention outside of current country standard of care.
Groups:
- Intervention Arm Stage 1: Annual universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care
  Adverse events monitored among persons initiating ART outside of National guidelines
- Intervention Arm Stage II: Baseline universal community-based HIV and multi-disease testing; ART eligibility for all HIV+; ART delivery using streamlined patient-centered care; targeted population-level PrEP
  Adverse events monitored among persons initiating PrEP
Arm/Group | Intervention Arm Stage 1 | Intervention Arm Stage II
All-Cause Mortality (participants affected / at risk) | 1217/79818 | 18/5447
Serious Adverse Events (participants affected / at risk) | 89/1671 | 50/5447
Other Adverse Events (participants affected / at risk) | 80/1671 | 17/5447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm Stage 1 (N=1671) | Intervention Arm Stage II (N=5447)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 13 (14) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cutaneous Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Diarrhea (General disorders) | 1 (1) | 0 (0)
Elevated ALT (Renal and urinary disorders) | 4 (4) | 0 (0)
Elevated AST (Renal and urinary disorders) | 2 (2) | 0 (0)
Elevated Creatinine (Renal and urinary disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Genital Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Intoxication (General disorders) | 1 (1) | 0 (0)
Neuromuscular weakness (Nervous system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 6 (7) | 1 (1)
Pre-term Labor (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Soft Tissue Injury (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 3 (3)
Temperature (General disorders) | 1 (1) | 0 (0)
Unintentional Weight Loss (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Urticaria (Renal and urinary disorders) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 2 (2) | 0 (0)
Vomiting (General disorders) | 3 (3) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wound (General disorders) | 1 (1) | 0 (0)
Fetal Demise (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Fever (General disorders) | 8 (8) | 0 (0)
Blood clot in brain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cesarean Infant Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Head Injury (Nervous system disorders) | 0 (0) | 1 (1)
Uterine Fibroids (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pulmonary Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ruptured Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Seroconversion (Infections and infestations) | 0 (0) | 25 (25)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Typhoid (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm Stage 1 (N=1671) | Intervention Arm Stage II (N=5447)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 4 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 18 (18) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Dizziness (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Eye Discharge (Eye disorders) | 1 (1) | 0 (0)
Elevated ALT (Renal and urinary disorders) | 11 (11) | 0 (0)
Elevated AST (Renal and urinary disorders) | 6 (6) | 0 (0)
Elevated Creatinine (Renal and urinary disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyponatraemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leucopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Renal and urinary disorders) | 11 (11) | 0 (0)
Pain (General disorders) | 6 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Spontaneous Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Thrombocytopenia (Renal and urinary disorders) | 4 (4) | 0 (0)
Unintentional Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 2 (2) | 0 (0)
Elevated Bilirubin (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Uterine Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4)
Dizzinesss (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In the second stage, following re-randomization, there was a DSMB approved study modification due to policy changes in standard of care. As a result, outcomes were only assessed among participants in the intervention arm who were offered PrEP. No data were collected in the control arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT01864603/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT01864603/SAP_001.pdf